CLINICAL TRIAL: NCT02754518
Title: Demonstration of Reverse Remodeling Effects of Entresto (Valsartan/Sacubitril) Using Echocardiography Endocardial Surface Analysis
Brief Title: Demonstration of Reverse Remodeling Effects of Entresto. Using Echocardiography Endocardial Surface Analysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB15-1410
Record Dates: First submitted 2016-04-22; First posted 2016-04-28 (Estimated); Results first posted 2021-01-29 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open label Entresto (Other): All subjects will take Entresto, a drug recently approved by the US Food and Drug Administration (FDA) for heart failure. In this study subjects will take this drug as they normally would for their standard of care.
  Interventions: Drug: Entresto

INTERVENTIONS:
Drug: Entresto
  Other Names: valsartan/sacubitril

SUMMARY:
This study intends to measure the effects of valsartan/sacubitril compared to baseline standard medical heart failure therapy on reverse remodeling using echocardiographic endocardial surface analysis techniques to assess changes in ventricular volume, function, and shape.

DETAILED DESCRIPTION:
This study intends to measure the effects of valsartan/sacubitril compared to baseline standard medical heart failure therapy on reverse remodeling using echocardiographic endocardial surface analysis techniques to assess changes in ventricular volume, function, and shape. Furthermore, Metaiodobenzylguanidine (MIBG) scintigraphy and the heart to mediastinum ratio will be used to assess Left Ventricle (LV) volume regression and risk reduction. The investigators also intend to measure the effects of valsartan/sacubitril on exercise capacity as assessed by the 6 minute walk test and peak Volume of Oxygen (V02) on cardiopulmonary exercise testing. Additionally, the investigators will examine the impact of valsartan/sacubitril on functional status and quality of life using the Kansas City Cardiomyopathy Questionnaire (KCCQ) and Qualia Health (a novel iPhone application that incorporates Fitbit technology to provide a "real time" daily 6 minute step count and assesses quality of life using a series of short targeted questions. The investigators will also measure Brain Natriuretic Peptide (BNP), N-terminal of the Prohormone Brain Natriuretic Peptide (NT-proBNP), and Rho-kinase (a biomarker associated with heart failure) levels at multiple time-points throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged ≥18 years
2. Congestive Heart Failure (CHF) New York Heart Association (NYHA) class II-IV with 25%≤ Left Ventricular Ejection Fraction (LVEF) ≤40% (ECHO within last 6 months)

   * NT-proBNP ≥ 600 pg/mL OR
   * NT-proBNP ≥ 400 pg/mL and a hospitalization for heart failure within the last 12 months
3. Stable and optimized on an angiotensin-converting-enzyme inhibitor (ACEI) equivalent to enalapril ≥ 10 twice a day (BID) for at least 4 weeks
4. Stable and optimized on a beta-blocker for at least 4 weeks
5. Optimized dosing of aldosterone antagonist at stable dose for at least 4 weeks

Exclusion Criteria:

1. History of angioedema
2. estimated glomerular filtration rate (eGFR) < 30 ml/min/1.73 m2 at screening
3. Serum potassium > 5.2 mmol/L at screening
4. Symptomatic hypotension as defined by Investigator, systolic blood pressure (SBP) < 100 mmHg at screening
5. Current acute decompensated heart failure
6. History of severe pulmonary disease
7. Active malignancy
8. Requirement for treatment with both angiotensin-converting-enzyme inhibitor (ACEI) and angiotensin receptor blockers (ARB)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Kalantari, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a prospective, single-arm longitudinal study, 40 patients were initiated on valsartan/sacubitril after a two week run in period of ACE or ARB alone.
Groups:
- Open Label Entresto: All subjects will take Entresto, a drug recently approved by the US Food and Drug Administration (FDA) for heart failure. In this study subjects will take this drug as they normally would for their standard of care.
  Entresto
Period: Overall Study
Arm/Group | Open Label Entresto
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Open Label Entresto
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Ethnicity: American Indian or Alaska Native | 0
  Ethnicity: Asian | 2
  Ethnicity: Native Hawaiian or Other Pacific Islander | 0
  Ethnicity: Black or African American | 23
  Ethnicity: White | 15
  Ethnicity: More than one race | 0
  Ethnicity: Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40
New York Heart Association (NYHA) Class [Count of Participants; unit: Participants] — New York Heart Association (NYHA) Functional Classification.
  I: No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, shortness of breath (SOB).
  II: Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, SOB.
  III: Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or SOB.
  IV: Unable to do any physical activity without discomfort. Symptoms of heart failure at rest.
  Participants
    Class II | 26
    Class III | 13
    Unknown | 1
Heart Failure Etiology [Count of Participants; unit: Participants]
  Ischemic (ICM) | 10
  Nonischemic (NICM) | 24
  Unknown | 6
LV Remodeling [Mean (Standard Deviation); unit: percent]
  LV Ejection Fraction | 32 (7)
  Conicity | 0.75 (0.03)
  Sphericity | 0.73 (0.05)
LV Remodeling-Global Longitudinal Strain (%) [Mean (Standard Deviation); unit: percent] | -12.9 (2.8)
LV Remodeling [Median (Inter-Quartile Range); unit: mL] — Population: Some patients have incomplete data.
  mL
    Left Atrial Volume | 90.9 [67.7 to 111.1]
    3D End-Diastolic Volume: number analyzed (Participants) | 39
    3D End-Diastolic Volume | 243.5 [190.1 to 302.1]
    3D End-Systolic Volume: number analyzed (Participants) | 39
    3D End-Systolic Volume | 159.7 [118.9 to 207.9]
LV Remodeling [Mean (Standard Deviation); unit: cm]
  2D End-Diastolic Diameter | 6.0 (0.8)
  2D End-Systolic Diameter | 5.3 (0.9)
RV Remodeling [Median (Inter-Quartile Range); unit: cm]
  End-Diastolic Volume | 143 [121 to 174]
  End Systolic Volume | 73 [51 to 97]
RV Remodeling [Mean (Standard Deviation); unit: percent]
  Ejection Fraction | 50 (10)
  Septal Curvature | 0.86 (0.15)
RV Remodeling - Free-Wall Curvature [Median (Inter-Quartile Range); unit: percent] | 1.17 [1.09 to 1.22]
RV Remodeling - Tricuspid Regurgitation [Count of Participants; unit: Participants]
  No | 3
  Trace | 30
  Mild | 4
  Mild-Moderate | 2
  Moderate | 0
  Moderate-Severe | 1
  Severe | 0
Exercise Performance- 6 Minute Walk [Mean (Standard Deviation); unit: Meter] | 425 (102)
Exercise Performance - CPX -Peak RER [Mean (Standard Deviation); unit: meters] | 1.14 (0.1)
Exercise Performance - CPX - Peak VO2 [Median (Inter-Quartile Range); unit: mL/kg/min] | 17.5 [13.7 to 22.4]
Exercise Performance - CPX - VE/VC02 [Median (Inter-Quartile Range); unit: ratio] | 33 [29 to 38]
Blood Pressure [Mean (Standard Deviation); unit: mmHg]
  Systolic | 127 (22.6)
  Diastolic | 76 (14.6)
Rho-kinase (Rock) [Median (Inter-Quartile Range); unit: ng/mL] | 1 [0.7 to 1.4]
hm ratio [Median (Inter-Quartile Range); unit: ratio] — Population: Some patients have incomplete data.
  ratio
    (MIBG) Early hm ratio: number analyzed (Participants) | 39
    (MIBG) Early hm ratio | 1.54 [1.34 to 1.61]
    (MIBG) Late hm ratio: number analyzed (Participants) | 39
    (MIBG) Late hm ratio | 1.43 [1.27 to 1.53]
NT-proBNP levels [Median (Inter-Quartile Range); unit: pg/mL] | 333 [130 to 1003]
Kansas City Cardiomyopathy Questionnaire (KCCQ) [Median (Inter-Quartile Range); unit: scores on a scale] — KCCQ is a 23-item instrument that is self-administered. KCCQ measures physical function, symptoms (specifically frequency, severity, and recent change), social function, self-efficacy and knowledge, and quality of life. Subscales and Total Score range from 0-100; higher scores show better health status.
  Developed and validated by Dr. John Spertus,MD of University of Missouri-Kansas City. Population: Clinical Summary Score is the sum of total symptom and physical function, and then rescaled to range from 0-100. Overall Summary Score is sum of total symptom, physical function, social limitations, and quality of life scores, and then rescaled to range from 0-100.
  Some patients had incomplete data.
  scores on a scale
    Physical limitation | 90 [71 to 100]
    Symptom Stability | 50 [50 to 50]
    Symptom Frequency | 89 [74 to 100]
    Symptom Burden | 92 [79 to 100]
    Total Symptom | 89 [71.5 to 100]
    Self Efficacy | 88 [75 to 100]
    Quality of Life Score | 67 [42 to 83]
    Social Limitation: number analyzed (Participants) | 39
    Social Limitation | 81 [56 to 94]
    Overall Summary | 82 [65 to 90]
    Clinical Summary | 91 [72 to 98]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in LV Remodeling 2D End-Diastolic Diameter (cm)
Description: LV Remodeling 2D End-Diastolic Diameter (cm)
Time Frame: Baseline,1 year
Population: All subjects will take Entresto, a drug recently approved by the US Food and Drug Administration (FDA) for heart failure.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Open Label Entresto
Number analyzed (Participants) | 40
cm
  Baseline | 6 (0.8)
  1 year: number analyzed (Participants) | 33
  1 year | 6 (0.7)
Statistical Analysis 1: Comparison: Open Label Entresto; Primary outcome was presented at baseline and 1-year as means +/- standard deviations based upon the Shapiro-Wilks test of normality, and then analyzed with paired t-tests; Test type: Other; p < 0.001, t-test, 2 sided — P-values are not adjusted for multiple comparisons. Tests were two-tailed, considered statistically significant with a p-value <0.05, and conducted using STATA MP version 15 (College Station, TX); Paired t-test

2. Primary Outcome: Change From Baseline in LV Remodeling 2D End-Systolic Diameter (cm)
Description: LV Remodeling 2D End-Systolic Diameter (cm)
Time Frame: Baseline,1 year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Open Label Entresto
Number analyzed (Participants) | 40
cm
  Baseline | 5.3 (0.9)
  1 year: number analyzed (Participants) | 33
  1 year | 4.5 (0.9)
Statistical Analysis 1: Comparison: Open Label Entresto; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; paired t-test

3. Primary Outcome: Change From Baseline in LV Remodeling Global Longitudinal Strain (%)
Description: LV Remodeling Global Longitudinal Strain (%)
Time Frame: Baseline,1 year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of global longitudinal strain
Arm/Group | Open Label Entresto
Number analyzed (Participants) | 40
percentage of global longitudinal strain
  Baseline | -12.9 (2.8)
  1 year: number analyzed (Participants) | 30
  1 year | -15.3 (3.5)
Statistical Analysis 1: Comparison: Open Label Entresto; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; paired t-test

4. Primary Outcome: Change From Baseline in LV Remodeling Left Atrial Volume (mL)
Description: LV Remodeling Left Atrial Volume (mL)
Time Frame: Baseline,1 year
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Open Label Entresto
Number analyzed (Participants) | 40
mL
  Baseline | 90.9 [67.7 to 111.1]
  1 year: number analyzed (Participants) | 32
  1 year | 65.6 [49.8 to 90.3]
Statistical Analysis 1: Comparison: Open Label Entresto; Primary outcome was presented at baseline and 1-year as medians (interquartile range) based upon the Shapiro-Wilks test of normality, and then analyzed with Wilcoxon signed-rank test; Test type: Other; p < 0.001, Sign test — [p-value comment as in outcome 1, analysis 1]

5. Primary Outcome: Change From Baseline in LV Remodeling 3D End-Diastolic Volume (mL)
Description: LV Remodeling 3D End-Diastolic Volume (mL)
Time Frame: Baseline,1 year
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Open Label Entresto
Number analyzed (Participants) | 39
mL
  Baseline | 243.5 [190.1 to 302.1]
  1 year: number analyzed (Participants) | 32
  1 year | 160.2 [118.8 to 214.8]
Statistical Analysis 1: Comparison: Open Label Entresto; [analysis description as in outcome 4, analysis 1]; Test type: Other; p < 0.001, Sign test — [p-value comment as in outcome 1, analysis 1]

6. Primary Outcome: Change From Baseline in LV Remodeling 3D End-Systolic Volume (mL)
Description: LV Remodeling 3D End-Systolic Volume (mL)
Time Frame: Baseline,1 year
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Open Label Entresto
Number analyzed (Participants) | 39
mL
  Baseline | 159.7 [118.9 to 207.9]
  1 year: number analyzed (Participants) | 32
  1 year | 90.7 [66.4 to 130.6]
Statistical Analysis 1: Comparison: Open Label Entresto; [analysis description as in outcome 4, analysis 1]; Test type: Other; p < 0.001, Sign test — [p-value comment as in outcome 1, analysis 1]

7. Primary Outcome: Change From Baseline in LV Remodeling LV Ejection Fraction (%)
Description: LV Remodeling LV Ejection Fraction (%)
Time Frame: Baseline,1 year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of ejection fraction
Arm/Group | Open Label Entresto
Number analyzed (Participants) | 40
percentage of ejection fraction
  Baseline | 32 (7)
  1 year: number analyzed (Participants) | 32
  1 year | 43 (9)
Statistical Analysis 1: Comparison: Open Label Entresto; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Paired t-test

8. Primary Outcome: Change From Baseline in LV Remodeling Conicity (%)
Description: LV Remodeling Conicity (%)
Time Frame: Baseline,1 year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of conicity
Arm/Group | Open Label Entresto
Number analyzed (Participants) | 40
percentage of conicity
  Baseline | 0.75 (0.03)
  1 year: number analyzed (Participants) | 11
  1 year | 0.77 (0.02)
Statistical Analysis 1: Comparison: Open Label Entresto; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.13, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; paired t-test

9. Primary Outcome: Change From Baseline in LV Remodeling Sphericity (%)
Description: LV Remodeling Sphericity (%)
Time Frame: Baseline,1 year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of sphericity
Arm/Group | Open Label Entresto
Number analyzed (Participants) | 40
percentage of sphericity
  Baseline | 0.73 (0.05)
  1 year: number analyzed (Participants) | 11
  1 year | 0.71 (0.03)
Statistical Analysis 1: Comparison: Open Label Entresto; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.95, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Paired t-test

10. Primary Outcome: Change From Baseline in RV Remodeling End-Diastolic Volume (mL)
Description: RV Remodeling End-Diastolic Volume (mL)
Time Frame: Baseline,1 year
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Open Label Entresto
Number analyzed (Participants) | 27
mL
  Baseline | 143 [121 to 174]
  1 year | 104 [83 to 145]
Statistical Analysis 1: Comparison: Open Label Entresto; [analysis description as in outcome 4, analysis 1]; Test type: Other; p < 0.001, Sign test — [p-value comment as in outcome 1, analysis 1]

11. Primary Outcome: Change From Baseline in RV Remodeling End Systolic Volume (mL)
Description: RV Remodeling End Systolic Volume (mL)
Time Frame: Baseline,1 year
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Open Label Entresto
Number analyzed (Participants) | 40
mL
  Baseline | 73 [51 to 97]
  1 year: number analyzed (Participants) | 27
  1 year | 47 [35.4 to 72.3]
Statistical Analysis 1: Comparison: Open Label Entresto; [analysis description as in outcome 4, analysis 1]; Test type: Other; p < 0.001, Sign test — [p-value comment as in outcome 1, analysis 1]

12. Primary Outcome: Change From Baseline in RV Remodeling Ejection Fraction (%)
Description: RV Remodeling Ejection Fraction (%)
Time Frame: Baseline,1 year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of ejection fraction
Arm/Group | Open Label Entresto
Number analyzed (Participants) | 40
percentage of ejection fraction
  Baseline | 50 (10)
  1 year: number analyzed (Participants) | 28
  1 year | 50 (8)
Statistical Analysis 1: Comparison: Open Label Entresto; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.65, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Paired T-test

13. Primary Outcome: Change From Baseline in RV Remodeling Septal Curvature (%)
Description: RV Remodeling Septal Curvature (%)
Time Frame: Baseline,1 year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of septal curvature
Arm/Group | Open Label Entresto
Number analyzed (Participants) | 40
percentage of septal curvature
  Baseline | 0.86 (0.15)
  1 year: number analyzed (Participants) | 9
  1 year | 0.77 (0.8)
Statistical Analysis 1: Comparison: Open Label Entresto; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.06, Sign test — [p-value comment as in outcome 1, analysis 1]

14. Primary Outcome: Change From Baseline in RV Remodeling Free-Wall Curvature (%)
Description: RV Remodeling Free-Wall Curvature (%)
Time Frame: Baseline,1 year
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of free-wall curvature
Arm/Group | Open Label Entresto
Number analyzed (Participants) | 40
percentage of free-wall curvature
  Baseline | 1.17 [1.09 to 1.22]
  1 year: number analyzed (Participants) | 9
  1 year | 1.14 [1.10 to 1.17]
Statistical Analysis 1: Comparison: Open Label Entresto; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.76, Sign test — [p-value comment as in outcome 1, analysis 1]

15. Primary Outcome: Change From Baseline in RV Remodeling Tricuspid Regurgitation
Description: RV Remodeling Tricuspid Regurgitation
Time Frame: Baseline,1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Entresto
Number analyzed (Participants) | 40
Participants
  Baseline: No | 3
  Baseline: Trace | 30
  Baseline: Mild | 4
  Baseline: Mild-Moderate | 2
  Baseline: Moderate | 0
  Baseline: Moderate-Severe | 1
  Baseline: Severe | 0
  1 year: number analyzed (Participants) | 33
  1 year: No | 8
  1 year: Trace | 16
  1 year: Mild | 9
  1 year: Mild-Moderate | 0
  1 year: Moderate | 0
  1 year: Moderate-Severe | 0
  1 year: Severe | 0
Statistical Analysis 1: Comparison: Open Label Entresto; Primary outcome was presented at baseline and 1-year as frequency and percentages based upon the Shapiro-Wilks test of normality, and then analyzed with the Fisher exact test; Test type: Other; p = 0.07, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

16. Secondary Outcome: Change From Baseline in Rho-associated Protein Kinase (ROCK)
Description: Rho-associated protein kinase (ROCK)
Time Frame: Baseline,1 year
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Open Label Entresto
Number analyzed (Participants) | 40
ng/mL
  Baseline | 1.1 [0.7 to 1.4]
  1 year: number analyzed (Participants) | 27
  1 year | 0.7 [0.5 to 1]
Statistical Analysis 1: Comparison: Open Label Entresto; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.001, Sign test — [p-value comment as in outcome 1, analysis 1]

17. Secondary Outcome: Change From Baseline in (MIBG) Early hm Ratio
Description: Cardiac 123Iodine-metaiodobenzylguanidine (MIBG) Early heart/mediastinum ratio (hm) ratio
Time Frame: Baseline,1 year
Population: All subjects will take Entresto, a drug recently approved by the US Food and Drug Administration (FDA) for heart failure.
  0 participants analyzed at 1 year as data were not collected.
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Open Label Entresto
Number analyzed (Participants) | 39
ratio
  Baseline | 1.54 [1.34 to 1.61]
  1 year: number analyzed (Participants) | 0

18. Secondary Outcome: Change From Baseline in (MIBG) Late hm Ratio
Description: Cardiac 123Iodine-metaiodobenzylguanidine (MIBG) Late heart/mediastinum ratio (hm) ratio
Time Frame: Baseline,1 year
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Open Label Entresto
Number analyzed (Participants) | 39
ratio
  Baseline | 1.43 [1.27 to 1.53]
  1 year: number analyzed (Participants) | 0

19. Secondary Outcome: Change From Baseline in NT-proBNP Levels
Description: NT-proBNP levels (pg/ml)
Time Frame: Baseline,1 year
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Open Label Entresto
Number analyzed (Participants) | 37
pg/ml
  Baseline | 333 [130 to 1003]
  1 year: number analyzed (Participants) | 31
  1 year | 290 [64 to 616]
Statistical Analysis 1: Comparison: Open Label Entresto; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.03, Sign test — [p-value comment as in outcome 1, analysis 1]

20. Secondary Outcome: Change From Baseline in Exercise Performance - 6 Minute Walk
Description: Exercise Performance - 6 Minute Walk
Time Frame: Baseline,1 year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Open Label Entresto
Number analyzed (Participants) | 40
meters
  Baseline | 425 (102)
  1 year: number analyzed (Participants) | 33
  1 year | 486 (124)
Statistical Analysis 1: Comparison: Open Label Entresto; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Paired t-test

21. Secondary Outcome: Change From Baseline in Exercise Performance - CPX - Peak VO2 (mL/kg/Min)
Description: Exercise Performance - CPX - Peak VO2 (mL/kg/min)
Time Frame: Baseline,1 year
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mL/kg/min
Arm/Group | Open Label Entresto
Number analyzed (Participants) | 40
mL/kg/min
  Baseline | 17.5 [13.7 to 22.4]
  1 year: number analyzed (Participants) | 31
  1 year | 19.5 [14.8 to 23]
Statistical Analysis 1: Comparison: Open Label Entresto; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.02, Sign test — [p-value comment as in outcome 1, analysis 1]

22. Secondary Outcome: Change From Baseline in Exercise Performance - CPX - Peak RER
Description: Exercise Performance - CPX - Peak RER (Respiratory Exchange Ratio)
Time Frame: Baseline,1 year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Open Label Entresto
Number analyzed (Participants) | 40
ratio
  Baseline | 1.14 (0.10)
  1 year: number analyzed (Participants) | 31
  1 year | 1.06 (0.10)
Statistical Analysis 1: Comparison: Open Label Entresto; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Paired t-test

23. Secondary Outcome: Change From Baseline in Exercise Performance - CPX - VE/VC02
Description: Exercise Performance - CPX - VE/VC02
Time Frame: Baseline,1 year
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Open Label Entresto
Number analyzed (Participants) | 40
ratio
  Baseline | 33 [29 to 38]
  1 year: number analyzed (Participants) | 30
  1 year | 33 [30 to 40]
Statistical Analysis 1: Comparison: Open Label Entresto; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.82, Sign test — [p-value comment as in outcome 1, analysis 1]

24. Secondary Outcome: Change From Baseline in Blood Pressure - Systolic (mmHg)
Description: Blood Pressure - Systolic (mmHg)
Time Frame: Baseline,1 year
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Open Label Entresto
Number analyzed (Participants) | 40
mmHg
  Baseline | 131 [122 to 143]
  1 year: number analyzed (Participants) | 35
  1 year | 114 [105 to 124]
Statistical Analysis 1: Comparison: Open Label Entresto; [analysis description as in outcome 4, analysis 1]; Test type: Other; p < 0.001, Sign test — [p-value comment as in outcome 1, analysis 1]

25. Secondary Outcome: Change From Baseline in Blood Pressure - Diastolic (mmHg)
Description: Blood Pressure - Diastolic (mmHg)
Time Frame: Baseline,1 year
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Open Label Entresto
Number analyzed (Participants) | 40
mmHg
  Baseline | 82 [74 to 89]
  1 year: number analyzed (Participants) | 35
  1 year | 76 [66 to 84]
Statistical Analysis 1: Comparison: Open Label Entresto; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.01, Sign test — [p-value comment as in outcome 1, analysis 1]

26. Secondary Outcome: Change From Baseline in KCCQ - Physical Limitation
Description: KCCQ is a 23-item instrument that is self-administered. KCCQ measures physical function, symptoms (specifically frequency, severity, and recent change), social function, self-efficacy and knowledge, and quality of life. Subscales and Total Score range from 0-100; higher scores show better health status.
  Developed and validated by Dr. John Spertus,MD of University of Missouri-Kansas City.
Time Frame: Baseline,1 year
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Open Label Entresto
Number analyzed (Participants) | 40
score on a scale
  Baseline | 90 [71 to 100]
  1 year: number analyzed (Participants) | 23
  1 year | 96 [88 to 100]
Statistical Analysis 1: Comparison: Open Label Entresto; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.11, Sign test — [p-value comment as in outcome 1, analysis 1]

27. Secondary Outcome: Change From Baseline in KCCQ - Symptom Stability
Description: as for outcome 26
Time Frame: Baseline,1 year
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Open Label Entresto
Number analyzed (Participants) | 40
score on a scale
  Baseline | 50 [50 to 50]
  1 year: number analyzed (Participants) | 24
  1 year | 50 [50 to 100]
Statistical Analysis 1: Comparison: Open Label Entresto; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.17, Sign test — [p-value comment as in outcome 1, analysis 1]

28. Secondary Outcome: Change From Baseline in KCCQ - Symptom Frequency
Description: as for outcome 26
Time Frame: Baseline,1 year
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Open Label Entresto
Number analyzed (Participants) | 40
score on a scale
  Baseline | 89 [74 to 100]
  1 year: number analyzed (Participants) | 24
  1 year | 92 [85 to 98]
Statistical Analysis 1: Comparison: Open Label Entresto; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.035, Sign test — [p-value comment as in outcome 1, analysis 1]

29. Secondary Outcome: Change From Baseline in KCCQ - Symptom Burden
Description: as for outcome 26
Time Frame: Baseline,1 year
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Open Label Entresto
Number analyzed (Participants) | 40
score on a scale
  Baseline | 92 [79 to 100]
  1 year: number analyzed (Participants) | 24
  1 year | 92 [83 to 100]
Statistical Analysis 1: Comparison: Open Label Entresto; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.059, Sign test — [p-value comment as in outcome 1, analysis 1]

30. Secondary Outcome: Change From Baseline in KCCQ - Total Symptom
Description: as for outcome 26
Time Frame: Baseline,1 year
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Open Label Entresto
Number analyzed (Participants) | 40
score on a scale
  Baseline | 89 [71.5 to 100]
  1 year: number analyzed (Participants) | 24
  1 year | 92 [86 to 99]
Statistical Analysis 1: Comparison: Open Label Entresto; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.054, Sign test — [p-value comment as in outcome 1, analysis 1]

31. Secondary Outcome: Change From Baseline in KCCQ - Self Efficacy
Description: as for outcome 26
Time Frame: Baseline,1 year
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Open Label Entresto
Number analyzed (Participants) | 40
score on a scale
  Baseline | 88 [75 to 100]
  1 year: number analyzed (Participants) | 24
  1 year | 100 [75 to 100]
Statistical Analysis 1: Comparison: Open Label Entresto; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.28, Sign test — [p-value comment as in outcome 1, analysis 1]

32. Secondary Outcome: Change From Baseline in KCCQ - Quality of Life Score
Description: as for outcome 26
Time Frame: Baseline,1 year
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Open Label Entresto
Number analyzed (Participants) | 40
score on a scale
  Baseline | 67 [42 to 83]
  1 year: number analyzed (Participants) | 24
  1 year | 83 [67 to 100]
Statistical Analysis 1: Comparison: Open Label Entresto; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.002, Sign test — [p-value comment as in outcome 1, analysis 1]

33. Secondary Outcome: Change From Baseline in KCCQ - Social Limitation
Description: as for outcome 26
Time Frame: Baseline,1 year
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Open Label Entresto
Number analyzed (Participants) | 39
score on a scale
  Baseline | 81 [56 to 94]
  1 year: number analyzed (Participants) | 24
  1 year | 94 [81 to 100]
Statistical Analysis 1: Comparison: Open Label Entresto; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.008, Sign test — [p-value comment as in outcome 1, analysis 1]

34. Secondary Outcome: Change From Baseline in KCCQ - Overall Summary
Description: as for outcome 26
Time Frame: Baseline,1 year
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Open Label Entresto
Number analyzed (Participants) | 40
score on a scale
  Baseline | 82 [65 to 90]
  1 year: number analyzed (Participants) | 24
  1 year | 90 [79.5 to 97.5]
Statistical Analysis 1: Comparison: Open Label Entresto; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.005, Sign test — [p-value comment as in outcome 1, analysis 1]

35. Secondary Outcome: Change From Baseline in KCCQ - Clinical Summary
Description: as for outcome 26
Time Frame: Baseline,1 year
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Open Label Entresto
Number analyzed (Participants) | 40
score on a scale
  Baseline | 91 [72 to 98]
  1 year: number analyzed (Participants) | 24
  1 year | 94.5 [87 to 98.5]
Statistical Analysis 1: Comparison: Open Label Entresto; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.056, Sign test — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Open Label Entresto: REMODEL is a prospective, single-arm longitudinal study investigating the structural, neurohormonal and functional effects of sacubitril/valsartan. Patients with New York Heart Association (NYHA) Class II-III HFrEF who were on optimal guideline directed medical therapy for at least three months with an LVEF between 20-40% who otherwise met inclusion and exclusion criteria similar to that of the Paradigm Trial were eligible for enrollment.
Arm/Group | Open Label Entresto
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 4/40
Other Adverse Events (participants affected / at risk) | 4/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Entresto (N=40)
Hypotension (Cardiac disorders) | 4 (4) — Hypotension
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Entresto (N=40)
Hypotension (Cardiac disorders) | 4 (40)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-25): https://cdn.clinicaltrials.gov/large-docs/18/NCT02754518/Prot_SAP_000.pdf